CLINICAL TRIAL: NCT01432522
Title: Comparison of Absorption of Epinephrine Into the Circulation After Epinephrine Intranasal Spray Administration and After Intramuscular Injection
Brief Title: A Study for Absorption of Intranasal Epinephrine Compared to Conventional Intramuscular Epinephrine
Acronym: Epinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Pakit Vichyanond, MD, Professor of Pediatrics, Siriraj Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 078/2550
Record Dates: First submitted 2011-01-19; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Anaphylaxis
Keywords: Intranasal epinephrine; Plasma epinephrine level
MeSH Terms: conditions — Anaphylaxis | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- epinephrine IN, epinephrine IM, saline IN (Experimental): 1. Intranasal saline
  2. Intramuscular epinephrine
  3. Intranasal epinephrine
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Epinephrine — 1. Intranasal epinephrine 5 mg /spray
  2. Intramuscular epinephrine 0.3 mg
  3. Intranasal saline spray
  Other Names: adrenaline

SUMMARY:
This study is a preliminary report of pharmacokinetic data of epinephrine administered via intranasal route (IN) comparing with intramuscular (IM) route in healthy adult volunteers.

DETAILED DESCRIPTION:
Patients are reluctant to use Epipen® on emergency basis, perhaps because of improperly training, hesitancy and fear of needle. Other route of administration of epinephrine (EPI) may be more benefit such as intranasal route.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects
2. 18-30 years-old

Exclusion Criteria:

1. Pregnancy
2. Subjected who use current medication that interfere with result of plasma epinephrine level such as pseudoephedrine

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics of epinephrine | predose, 5 , 10, 15, 20, 30, 45, 60, 90, 120, 180 minutes post-dose
  Cmax, Area Under Curve, Tmax of epinephrine compare between 0.3 mg intramuscular and 5 mg intranasal route

SECONDARY OUTCOMES:
Numbers of participants with adverse events as a measure of safety and tolerability | 1 year
  Any side effects from such administration such as bad smelling, sorethroat.

CONTACTS AND LOCATIONS:
Overall Officials: Pakit Vichyanond, MD., Study Director — Siriraj medical school, Mahidol Univrsity
Locations (1):
- Facaulty of Medicine, Siriraj Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Simons FE, Gu X, Simons KJ. Epinephrine absorption in adults: intramuscular versus subcutaneous injection. J Allergy Clin Immunol. 2001 Nov;108(5):871-3. doi: 10.1067/mai.2001.119409. PMID 11692118
- [Result] Rawas-Qalaji MM, Simons FE, Simons KJ. Sublingual epinephrine tablets versus intramuscular injection of epinephrine: dose equivalence for potential treatment of anaphylaxis. J Allergy Clin Immunol. 2006 Feb;117(2):398-403. doi: 10.1016/j.jaci.2005.12.1310. PMID 16461140
- [Result] Simons FE, Gu X, Johnston LM, Simons KJ. Can epinephrine inhalations be substituted for epinephrine injection in children at risk for systemic anaphylaxis? Pediatrics. 2000 Nov;106(5):1040-4. doi: 10.1542/peds.106.5.1040. PMID 11061773
- [Result] Heilborn H, Hjemdahl P, Daleskog M, Adamsson U. Comparison of subcutaneous injection and high-dose inhalation of epinephrine--implications for self-treatment to prevent anaphylaxis. J Allergy Clin Immunol. 1986 Dec;78(6):1174-9. doi: 10.1016/0091-6749(86)90268-x. PMID 3782679